CLINICAL TRIAL: NCT03893747
Title: Three Batches Consistency, Immunity Duration and Safety of Inactivated Enterovirus 71 Vaccine Post-marketing Among Children Aged 6-35 Months in China
Brief Title: Immunity and Safety of Inactivated Enterovirus 71 Vaccine Post-marketing Among Children Aged 6-35 Months in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Wuhan Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT048-2
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- the first batch vaccine producted by 40 L reactor (Experimental): 500 subjects will be randomly received the first batch vaccine producted by 40 L reactor
  Interventions: Biological: The first batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor
- the second batch vaccine producted by 40 L reactor (Experimental): 500 subjects will be randomly received the second batch vaccine producted by 40 L reactor
  Interventions: Biological: The second batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor
- the third batch vaccine producted by 40 L reactor (Experimental): 500 subjects will be randomly received the third batch vaccine producted by 40 L reactor
  Interventions: Biological: The third batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor
- the first batch vaccine producted by 150 L reactor (Experimental): 500 subjects will be randomly received the first batch vaccine producted by 150 L reactor
  Interventions: Biological: The first batch of inactivated EV-A71 vaccine (vero cell) producted by 150 L reactor
- the second batch vaccine producted by 150 L reactor (Experimental): 500 subjects will be randomly received the second batch vaccine producted by 150 L reactor
  Interventions: Biological: The second batch of inactivated EV-A71 vaccine (vero cell) producted by 150 L reactor
- the third batch vaccine proudected by 150 L reactor (Experimental): 500 subjects will be randomly received the third batch vaccine producted by 150 L reactor
  Interventions: Biological: The third batch of inactivated EV-A71 vaccine (vero cell) proudected by 150 L reactor

INTERVENTIONS:
Biological: The first batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor — 500 subjects will be randomized to receive the first batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor
  Arms: the first batch vaccine producted by 40 L reactor
Biological: The second batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor — 500 subjects will be randomized to receive the second batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor
  Arms: the second batch vaccine producted by 40 L reactor
Biological: The third batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor — 500 subjects will be randomized to receive the third batch of inactivated EV-A71 vaccine (vero cell) producted by 40 L reactor
  Arms: the third batch vaccine producted by 40 L reactor
Biological: The first batch of inactivated EV-A71 vaccine (vero cell) producted by 150 L reactor — 500 subjects will be randomized to receive the first batch of inactivated EV-A71 vaccine (vero cell) producted by 150 L reactor
  Arms: the first batch vaccine producted by 150 L reactor
Biological: The second batch of inactivated EV-A71 vaccine (vero cell) producted by 150 L reactor — 500 subjects will be randomized to receive the second batch of inactivated EV-A71 vaccine (vero cell) producted by 150 L reactor
  Arms: the second batch vaccine producted by 150 L reactor
Biological: The third batch of inactivated EV-A71 vaccine (vero cell) proudected by 150 L reactor — 500 subjects will be randomized to receive the third batch of inactivated EV-A71 vaccine (vero cell) proudected by 150 L reactor
  Arms: the third batch vaccine proudected by 150 L reactor

SUMMARY:
This study evaluates three batches consistency, immunity duration and safety of inactivated Enterovirus 71(EV-A71) vaccine(vero cell) post-marketing among children aged 6-35months in China.3000 subjects will be recruited in this study, of who 1500 subjects will be randomly assigned in a ratio of 1:1:1 to receive one of the three batches of EV-A71 vaccines manufactured by 40L capacity reactor, other 1500 subjects will be randomly assigned in a ratio of 1:1:1 to receive one of the three batches of EV-A71 vaccines manufactured by 150L capacity reactor. Vaccine wil be administrated according to a two doses of schedule given at day 0 and 28. Sample will be collected at day 0, day 56 and at month 13 after vaccinaiton.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6-35 months
* Subjects who have been clinically judged to be healthy by the researcher after being asked about the medical history and related physical examination
* The subjects' guardians agree the requirements of the protocol and the relevant follow up visits
* The subjects' guardians agree and sign the informed consent
* Subjects who have no relocation or long-term travel plan within one year and are able to comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

* Subject who has a medical history of HFMD caused by EV71 or has been vaccinated with EV71 vaccine
* Subject that has a history of allergies to vaccines or vaccine ingredients, and has serious side effects on vaccines, such as allergies, urticaria, dyspnea, vascular neuroedema or abdominal pain
* Subject who has congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Subject who has a history of epilepsy, convulsion or convulsion, or a family history of mental illness
* Subject who has autoimmune disease or immune deficiency, or whose parents and siblings have autoimmune disease or immune deficiency
* Subject who has a history of asthma, vascular and neuroedema, diabetes or malignant tumor
* Subject who has a thyroid resection history, or received treatment due to thyroid disease in the past 12 months
* Subject who has an abnormal coagulation function (such as coagulation factor deficiency, coagulant disease, platelet abnormality) or obvious bruising or clotting disorder which was diagnosed by doctors.
* Asplenia, functional asplenia, or splenectomy due to any circumstances
* Acute onset of various acute or chronic diseases in the last 7 days
* Immunosuppressant therapy, antiallergic therapy, cytotoxicity therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, surface corticosteroid therapy for acute non-dermatitis) in the past 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicines or vaccines in last 1 month
* Any prior administration of attenuated live vaccine in last 15 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Under the anti-TB prevention or therapy
* Underarm temperature > 37.0 ℃ for fever before vaccination
* Other factors that are not suitable for clinical trials according to the judgment of researchers

Exclusion Criteria for the second dose:

* Have severe allergic reaction after first dose
* Have severe adverse reactions related to first dose
* Any situation meet the exclusion criteria stated in the exclusion criteria for first dose
* Acute infection or illness
* Other factors that are not suitable for clinical trials according to the judgment of researchers

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Consistency of different batches for geometric mean titre(GMT) after vaccination | 56 days after vaccination
  Consistency of different batches for GMT of EV-A71 neutralizing antibody on 56 day after vaccination
Incidence and severity of adverse reactions/adverse events after each dose | 1 month after each dose
  Incidence and severity of adverse reactions/adverse events within 1 month after each dose

SECONDARY OUTCOMES:
Incidence of sever adverse events after vaccination | 13 months after vaccination
  Incidence of sever adverse events within 13 months after vaccination
GMTof EV-A71 neutralizing antibody on day 56 after vaccination | 56 days after vaccination
  GMTof EV-A71 neutralizing antibody on day 56 after vaccination for different batchs
Positive rate of EV-A71 neutralizing antibody on day 56 after vaccination | 56 days after vaccination
  Positive rate of EV-A71 neutralizing antibody on day 56 after vaccination for different batchs
Seroconversion rate of EV-A71 neutralizing antibody on day 56 after vaccination | 56 days after vaccination
  Seroconversion rate of EV-A71 neutralizing antibody on day 56 after vaccination for different batchs
Geometric Mean Fold Increase(GMFI) of EV-A71 neutralizing antibody on day 56 after vaccination | 56 days after vaccination
  Geometric Mean Fold Increase(GMFI) of EV-A71 neutralizing antibody on day 56 after vaccination for different batchs
GMTof EV-A71 neutralizing antibody on month 13 after vaccination | 13 months after vaccination
  GMTof EV-A71 neutralizing antibody on month 13 after vaccination for different batchs
Positive rate of EV-A71 neutralizing antibody on month 13 after vaccination | 13 months after vaccination
  Positive rate of EV-A71 neutralizing antibody on month 13 after vaccination for different batchs

CONTACTS AND LOCATIONS:
Locations (1):
- Fengcai Zhu, Nanjing, China